CLINICAL TRIAL: NCT00178945
Title: Randomized, Double-Blind, Placebo-Controlled, Crossover Study of Botulinum Toxin Type A (Botox) for the Treatment of Pain Associated With Cervical Dystonia and Refractory Cervicothoracic Myofascial Pain Syndrome
Brief Title: Botulinum Toxin Type A (Botox) for the Treatment of Cervical Dystonia and Upper Thoracic Muscular Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Thomas L Davis, Dr. Thomas L. Davis, Vanderbilt University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 030797
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2007-08

CONDITIONS: Refractory Cervicothoracic Myofascial Pain Syndrome (CMPS); Cervical Dystonia
MeSH Terms: conditions — Torticollis | interventions — Botulinum Toxins, Type A

INTERVENTIONS:
Drug: Botulinum Toxin Type A

SUMMARY:
The purpose of this study is to investigate the use of injections of Botox (botulinum toxin type A) for the treatment of chronic neck pain. Botox is an approved treatment for patients with cervical dystonia. Cervical dystonia is a chronic condition characterized by involuntary movements of the neck that are often painful. In this study, the response from Botox in patients with neck pain not associated with cervical dystonia will be compared to the pain response in patients with cervical dystonia.

DETAILED DESCRIPTION:
Cervical dystonia (CD) is a condition characterized by involuntary movements of the neck. Generally these movements are rotational and are frequently associated with significant pain. Treatment of CD with oral medications is usually unsuccessful and the current treatment of choice for the majority of patients consists of periodic injections of botulinum toxin into the offending muscles. Resistant cases are considered candidates for selective surgical denervation procedures.

Botulinum toxin type A (Botox®) is a FDA approved treatment for CD. Botox® has been safely used to treat CD in our clinic since 1989. In controlled trials, Botox® significantly improved pain in patients with CD.

Cervico-thoracic pain syndromes not associated with dystonia (refractory cervicothoracic myofascial pain syndrome or CMPS) is a chronic regional pain syndrome. It is a common component in acute and chronic pain syndromes, occurring in up to 14% of the U.S. population. This pain is often resistant to treatment and is characterized by a series of tender trigger points. These are often injected with local anesthetics that provide temporary relief of pain in some patients. Recent uncontrolled trials have suggested that Botox® may be helpful in patients with CMPS. Most attempts to use Botox® to treat these Patients have utilized smaller doses of Botox® than those used typically to treat CD. Also, most studies have used Botox® injection into tender trigger points rather than into the belly of the muscle as is commonly done to treat CD.

In this study we will use doses of Botox® that are typically used to treat CD. Injections of Botox® will be guided by EMG to determine areas of involuntarily firing muscle rather than solely into tender trigger points. The results in patients with CMPS will be compared to the pain relief experienced with those with CD. It is hoped that this trial will provide pilot data for planning a larger safety and efficacy trial of Botox® for chronic cervico-thoracic pain not associated with CD.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient, male and female subjects, of any race, between 18 years of age and older. Female subjects of childbearing potential must have a negative urine pregnancy test result at the Screening/Baseline Visit. (A female is considered of childbearing potential unless she is postmenopausal or without a uterus and/or both ovaries.)
* Subjects suffering from cervicothoracic muscle pain with or without cervical dystonia. The pain must be of at least 3 months duration and characterized by a numerical pain rating score of at least 5 on the pain subscale of the TWSTR scale.
* Subjects who are able to understand the requirements of the study and sign an Informed Consent Form.

Exclusion Criteria:

* Female subjects who are pregnant (positive urine pregnancy test) or who have an infant they are breast-feeding or who are of childbearing potential and not practicing a reliable method of birth control (OCP or barrier).
* Subjects who have had standard trigger point injections with local anesthetics in the last 3 months.
* Subjects who have had chiropractic manipulation of the neck or upper thoracic region in the last 3 months or plan on having such manipulations during the study.
* Subjects, who by clinical evaluation and / or MRI study, are considered to have symptomatic cervical and/or thoracic disc pathology as primary etiology of their pain.
* Subjects whose cervical spine ROM is restricted in the setting of arthritic conditions (advanced osteoporosis, degenerative arthritis, ankylosing spondylitis).
* Significant medical or psychiatric comorbid disease, as deemed by the investigators
* Litigation involving the existence or cause for neck pain and/or headache
* Pending disability assessment
* Subjects with a diagnosis of Myasthenia Gravis, Eaton-Lambert Syndrome, Amyotrophic Lateral Sclerosis or any other disease that might interfere with neuromuscular function.
* Subjects currently using aminoglycoside antibiotics or agents that interfere with neuromuscular function.
* Subjects with profound atrophy or excessive weakness of the muscles in the target area(s) of injection.
* Subjects with an infection at the injection site or systemic infection (in this case, postpone study entry until one week following recovery).
* Subjects with an allergy or sensitivity to any component of the test medication.
* Subjects with a history of poor cooperation, non-compliance with medical treatment, or unreliability.
* Subjects currently participating in an investigational drug study or who have participated in an investigational drug study within 30 days of the Baseline Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2004-03; Study Completion 2006-03

PRIMARY OUTCOMES:
Score on the Pain Subscale of the TWSTRS

SECONDARY OUTCOMES:
Daily pain diary for 14 days post-injection
Safety profile at study exit

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L Davis, MD, Principal Investigator — Vanderbilt University Department of Neurology
Locations (1):
- Vanderbilt Department of Neurology, Nashville, Tennessee, United States

REFERENCES:
- [Background] Comella CL, Buchman AS, Tanner CM, Brown-Toms NC, Goetz CG. Botulinum toxin injection for spasmodic torticollis: increased magnitude of benefit with electromyographic assistance. Neurology. 1992 Apr;42(4):878-82. doi: 10.1212/wnl.42.4.878. PMID 1565246
- [Background] Freund BJ, Schwartz M. Treatment of whiplash associated neck pain [corrected] with botulinum toxin-A: a pilot study. J Rheumatol. 2000 Feb;27(2):481-4. PMID 10685817
- [Background] Gobel H, Heinze A, Heinze-Kuhn K, Austermann K. Botulinum toxin A in the treatment of headache syndromes and pericranial pain syndromes. Pain. 2001 Apr;91(3):195-199. doi: 10.1016/S0304-3959(01)00292-5. No abstract available. PMID 11275374
- [Background] Porta M. A comparative trial of botulinum toxin type A and methylprednisolone for the treatment of myofascial pain syndrome and pain from chronic muscle spasm. Pain. 2000 Mar;85(1-2):101-5. doi: 10.1016/s0304-3959(99)00264-x. PMID 10692608
- [Background] Wheeler AH, Goolkasian P, Gretz SS. A randomized, double-blind, prospective pilot study of botulinum toxin injection for refractory, unilateral, cervicothoracic, paraspinal, myofascial pain syndrome. Spine (Phila Pa 1976). 1998 Aug 1;23(15):1662-6; discussion 1667. doi: 10.1097/00007632-199808010-00009. PMID 9704373
- [Background] Wheeler AH, Goolkasian P, Gretz SS. Botulinum toxin A for the treatment of chronic neck pain. Pain. 2001 Dec;94(3):255-260. doi: 10.1016/S0304-3959(01)00358-X. PMID 11731062
- [Background] Botox(R) (Botulinum Toxin Type A) Purified Neurotoxin Complex. Package Insert.